CLINICAL TRIAL: NCT02888210
Title: Open Label, Phase/3 Study Assessing Safety and Efficacy of MD-15 Intraocular Lens in Patients With Aphakic Eye After Cataract Surgery
Brief Title: A Study Assessing Safety and Efficacy of MD-15 Intraocular Lens in Patients With Aphakic Eye After Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD151508
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MD-15 (Experimental): Investigational intraocular lens
  Interventions: Device: MD-15 Intraocular Lens

INTERVENTIONS:
Device: MD-15 Intraocular Lens

SUMMARY:
To evaluate safety and efficacy of MD-15 intraocular lens implanted into the aphakic eyes

ELIGIBILITY:
Inclusion Criteria:

* Patients who intend to undergo phacoemulsification cataract extraction

Exclusion Criteria:

* Patients who undergo secondary implantation
* Patients with vision loss induced by causes other than cataract
* Patients who the principal investigator/subinvestigator considers ineligible for enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-09-03 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
Corrected visual acuity | Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan